CLINICAL TRIAL: NCT03857022
Title: An Open-label Study to Evaluate the Effects of Enhanced External Counterpulsation on Tapering Inotropic Agents, Reduction of Brain Natriuretic Peptide and Rehospitalization in Patients With Heart Failure
Brief Title: A Study to Evaluate the Effects of EECP in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201805058DIPA
Record Dates: First submitted 2018-11-22; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: EECP, Heart Failure, NT-proBNP, Inotropic Agents
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Subjects of Heart failure with 'Enhanced External Counterpulsation" therapy
  Interventions: Device: Enhanced External Counterpulsa
- No 'Enhanced External Counterpulsation" (No Intervention): Subjects of Heart failure without 'Enhanced External Counterpulsation" therapy

INTERVENTIONS:
Device: Enhanced External Counterpulsa — The EECP therapy was given as a 1-hour session, once daily, for a total of 35 sessions. The daily urine amount, blood pressure, time for taper off positive inotropic agents, length of hospital stay, and will be monitored daily in the hospital stay. Patients will be followed-up if he or she can be released from hospital and the mortality, readmission for heart failure, and 6-minute walking distance will be checked at the end of 6th month. Plasma natriuretic peptide (BNP) or N-terminal pro-brain natriuretic peptide (NT-pro-BNP) levels will be checked at enrollment, day 35, and 6th month.
  Other Names: EECP
  Arms: Enhanced External Counterpulsation

SUMMARY:
The aims of this proposal are to investigate whether external enhanced counterpulsation (EECP) can facilitate heart failure (HF) patient weaning from intravenous infusion of positive inotropic agent, and thus decrease the length of hospital stay. The major adverse cardiovascular event (MACE) rate, including death and hospitalization for heart failure, will be monitored for 6 months if patients can be released from hospital. Exercise tolerance (6-minute walking distance) and plasma brain natriuretic peptide (BNP) level will be checked at the end of 6th month.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) patients dependent on intravenous infusion of positive inotropic agents have not only high mortality rate but also high morbidity in the prolonged hospital course. Medications such as angiotensin conversion enzyme inhibitor or angiotensin II receptor blocker may improve the survival of CHF patients. However, their implication is limited by the presence of hypotension secondary to low cardiac output. External enhanced counterpulsation (EECP), which generates the arterial and intracoronary hemodynamics similar to those of the intra-aortic balloon pump, is a recently approved treatment modality for patients with angina and heart failure. It can improve exercise capacity, quality of life and functional status.

Forty patients of (1) impaired left ventricular systolic function (LVEF 40%) and are dependent on intravenous infusion of positive inotropic agents but (2) without significant aortic regurgitation, overt fluid overload, or symptomatic peripheral arterial insufficiency will be included. They will be randomly allocated into EECP or control groups (n=20 for each). The EECP therapy was given as a 1-hour session, once daily, for a total of 35 sessions. The daily urine amount, blood pressure, time for taper off positive inotropic agents, length of hospital stay, and will be monitored daily in the hospital stay. Patients will be followed-up if he or she can be released from hospital and the mortality, readmission for heart failure, and 6-minute walking distance will be checked at the end of 6th month. Plasma natriuretic peptide (BNP) levels will be checked at enrollment, day 35, and 6th month.

ELIGIBILITY:
Inclusion criteria All answers must be "Yes" for study entry.

1. Male or female patients between 21-80 years of age.
2. Patients who have documented evidence of HF.

Evidence of HF required at least one of the following:

LVEF <40%. As assessed with 3 months prior to enrollment, and LVEF can be measured through echocardiogram or radionuclide angiocardiography (RNA); Clinical symptoms of HF, namely the presence of 2 major criteria or 1 major criterion + 2 minor criteria according to the Framingham score; NYHA Fc III or IV ACC/AHA stage D 3. Treated with inotropic agents. Inotropic agents include dopamine, dobutamine, milrinone, norepinephrine. Low dose is included as well. 4. Patients who sign the informed consent . Exclusion criteria All answers must be "No" for study entry.

1. Patients who had MI or coronary artery bypass grafting (CABG) within three months prior to the initiation of EECP treatment.
2. Patients who had transcatheter intervention (PCI) within 2 weeks prior to the initiation of EECP treatment.
3. Significant valvular heart disease, acute myocarditis.
4. Uncontrolled hypertension (blood pressure 180/100 mmHg).
5. Permanent pacemakers or implantable cardioverter defibrillators.
6. Non bypassed left main coronary with a luminal stenosis greater than 50%.
7. Severe symptomatic peripheral vascular disease.
8. History of deep vein thrombosis.
9. Phlebitis or stasis ulcer.
10. Bleeding diathesis, warfarin use with International Normalized Ratio 2.0.
11. Arial fibrillation or frequent ventricular premature beats that interferes with enhanced external counterpulsation triggering.
12. Baseline ECG abnormalities that would interfere with interpretation of exercise ECG.
13. Pregnant women, or women of childbearing potential but not using adequate birth control.
14. Any medical, psychological, cognitive, social or legal condition that would interfere with the ability of patient to give an Informed Consent and/or his or her capacity to comply with all study requirements, including the necessary time commitment.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
the natriuretic peptide (NT-pro-BNP) level will be reduced. | 7 week
  the natriuretic peptide (NT-pro-BNP) level will be reduced

SECONDARY OUTCOMES:
Weaning from intravenous infusion of positive inotropic agent | 24 week
  Weaning from intravenous infusion of positive inotropic agent
Decrease the length of hospital stay. | 24 week
  Decrease the length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Ming Lee, PhD, Principal Investigator — National Taiwan Unerversity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan